CLINICAL TRIAL: NCT07149012
Title: Artificial Intelligence for Surgical Care in War-Torn Sudan: Feasibility, Barriers, and Ethical Perspectives From a Conflict Zone
Brief Title: Artificial Intelligence for Surgical Care in War-Torn Sudan: Feasibility, Barriers, and Ethical Perspectives
Status: Completed | Type: Observational
Sponsor: Sudan Medical Specialization Board (Other Government)
Responsible Party: Principal Investigator, Alsadig Suliman, Principal Investigator, Sudan Medical Specialization Board
Other Study IDs: SMSB-AI-SURG-SUDAN-2025
Record Dates: First submitted 2025-08-15; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Surgical Procedures, Operative; Artificial Intelligence (AI); War Injury; Wounds and Injuries; Disasters; Health Services Accessibility; Developing Countries
Keywords: Artificial Intelligence; Surgeon Training; Technology Adoption in Surgery; Humanitarian Health
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Artificial Intelligence Awareness and Feasibility Assessment — A sequential explanatory mixed-methods assessment of surgeons' awareness, readiness, and perceived barriers to adopting artificial intelligence in surgical care during the ongoing Sudan conflict. The intervention consisted of:
  A validated, structured online questionnaire adapted from established AI awareness tools, assessing familiarity, perceived benefits, barriers, and ethical concerns.
  Semi-structured interviews with senior surgical residents and consultants to explore contextual and ethical perspectives in greater depth.
  The study did not implement AI tools in practice but focused on measuring feasibility and identifying requirements for future AI deployment in conflict-affected surgical systems.
  Other Names: AI Readiness Survey; AI in Surgical Care Study Sudan; AI Training and Barriers Assessment

SUMMARY:
This study is designed to examine how artificial intelligence (AI) could be applied to support surgical care in Sudan during the ongoing armed conflict. The conflict has disrupted hospital operations, displaced surgical teams, and limited access to specialists and modern technology. The investigators are conducting a survey of Sudanese surgeons working in public, private, military, and conflict-zone hospitals to assess awareness of AI, interest in its application, and perceived challenges. In addition, in-depth interviews with senior surgeons and residents are being performed to further explore perspectives on AI in surgical care.

This study represents one of the first attempts to investigate the role of AI in surgery within an active conflict setting in Africa. Findings from this research are expected to inform the design of AI tools that are tailored for fragile health systems, including offline and low-bandwidth environments.

ELIGIBILITY:
Inclusion Criteria:

* Sudanese general surgery residents or consultants.
* Currently working in public, private, military, NGO, or conflict-zone hospitals within Sudan.
* Able to provide informed consent.

Exclusion Criteria:

* Surgeons working outside Sudan.
* Non-surgical medical specialties.
* Inability or unwillingness to complete the survey or participate in interviews.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General surgery residents and consultants practicing in Sudan during the ongoing armed conflict, representing public, private, military, NGO, and conflict-zone hospitals across multiple regions. Participants include surgeons at various training levels, from early-year residents to senior consultants.
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Awareness of Artificial Intelligence in Surgical Care Among Sudanese Surgeons | At survey completion (October 2024 - June 2025)
  Measured using a structured questionnaire including domains of familiarity with AI concepts, perceived benefits, and potential applications in perioperative care. Responses are recorded on a 5-point Likert scale ranging from 1 (not at all familiar/beneficial/applicable) to 5 (very familiar/beneficial/applicable). Higher scores indicate greater awareness and more positive perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Alsadig Suliman, MBBS, Msc, Principal Investigator — Sudan Medical Specialization Board
Locations (1):
- Sudan Medical Specialization Board, Wad Medani, Al Jazirah, Sudan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive information collected from healthcare professionals working in conflict-affected regions. Sharing could risk identification of participants despite anonymization, given the small and specialized population.

REFERENCES:
- [Background] Alsaedi AR, Alneami N, Almajnoni F, Alamri O, Aljohni K, Alrwaily MK, Eid M, Budayr A, Alrehaili MA, Alghamdi MM, Almutairi ED, Eid MH. Perceived Worries in the Adoption of Artificial Intelligence Among Healthcare Professionals in Saudi Arabia: A Cross-Sectional Survey Study. Nurs Rep. 2024 Nov 28;14(4):3706-3721. doi: 10.3390/nursrep14040271. PMID 39728632
- [Background] Fleming CA, Ali O, Clements JM, Hirniak J, King M, Mohan HM, Nally DM, Burke J; Association of Surgeons in Training (ASIT). Surgical trainee experience and opinion of robotic surgery in surgical training and vision for the future: a snapshot study of pan-specialty surgical trainees. J Robot Surg. 2022 Oct;16(5):1073-1082. doi: 10.1007/s11701-021-01344-y. Epub 2021 Nov 26. PMID 34826106
- [Background] De Simone B, Abu-Zidan FM, Gumbs AA, Chouillard E, Di Saverio S, Sartelli M, Coccolini F, Ansaloni L, Collins T, Kluger Y, Moore EE, Litvin A, Leppaniemi A, Mascagni P, Milone L, Piccoli M, Abu-Hilal M, Sugrue M, Biffl WL, Catena F. Knowledge, attitude, and practice of artificial intelligence in emergency and trauma surgery, the ARIES project: an international web-based survey. World J Emerg Surg. 2022 Feb 10;17(1):10. doi: 10.1186/s13017-022-00413-3. PMID 35144645